CLINICAL TRIAL: NCT00428675
Title: Development of a Rapid Assessment Tool for Fatigue in Palliative Care
Brief Title: A New Tool for Assessing Fatigue in Individuals With Advanced Cancer
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: G118160539
Record Dates: First submitted 2007-01-26; First posted 2007-01-30 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2020-03

CONDITIONS: Neoplasms
Keywords: screening; fatigue
MeSH Terms: conditions — Neoplasms; Fatigue

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACI Instrument: 228 individuals completed the ACI instrument and other tools
  Interventions: Other: ACI instrument

INTERVENTIONS:
Other: ACI instrument — Following ethics approval, 17 experts in symptom management assisted with content validation during the pilot phase. In the main study, participants complete the FACT-F, the POMS-Vsf, and the ACI Instrument. A research assistant collected demographic information and assigned an ECOG score.

SUMMARY:
Fatigue is a common problem in advanced cancer and palliative care. The development of tools to measure fatigue, however, has been slowed by their inability to distinguish between fatigue and other related symptoms, such as tiredness. Our work suggests that these distinctions are important because they serve as markers for stressors associated with advancing disease. We have developed a tool that we believe will distinguish between these two states as well as exhaustion. In this study we will conduct some initial tests of this tool in preparation for its use as an outcome indicator in future studies.

DETAILED DESCRIPTION:
Based on a series of qualitative studies, our group is developing a new rapid fatigue assessment screening tool (rFAST) for use with individuals who have advanced cancer and are receiving care in either an active treatment or palliative setting.

Hypotheses:

1. The three tools (tiredness, fatigue, and exhaustion) in the rFAST are each defined by the same six dimensions: decline in stamina, decline in cognition, decline in sleep quality, diminished social network, and increased emotional reactivity
2. The five subscales of the tiredness, fatigue, and exhaustion scales are internally consistent.
3. Tiredness, fatigue, and exhaustion are distinct states that are manifested by unique patterns of scores on their 6 subscales
4. The mean POMS-Vsf scores of individuals who meet the definition of fatigue will be lower than the mean POMS-Vsf scores of individuals who meet the definition of tiredness and higher than the mean POMS-Vsf scores of individuals who meet the definition of exhaustion.

Objectives

1. To examine the factor structure of the tiredness, fatigue, and exhaustion scales of the rFAST.
2. To examine the internal consistency of the 5 subscales within the tired, fatigue, and exhaustion scales.
3. To compare actual rFAST scale scores to hypothesized scale profiles for tiredness, fatigue, and exhaustion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced cancer currently receiving treatment for either hematologic or lung cancer at the Jewish General Hospital in Montreal, or patients with advanced cancer currently receiving care through the Alberta Cancer Board (Cross Cancer Institute or Tom Baker Cancer Centre), or the palliative care programs associated with the regional health authority in Edmonton, Alberta who are at least 18 years old, able to read and write English, have a Folstein Mini Mental Status Exam score of at least 22.

Exclusion Criteria:

* Patients unable to give informed consent in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with advanced cancer
Sampling Method: Non-Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2005-10; Primary Completion 2007-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
ACI score | day 1
  Adaptive Capacity Index Score

CONTACTS AND LOCATIONS:
Overall Officials: Karin L Olson, Ph.D., Principal Investigator — University of Alberta
Locations (1):
- Faculty of Nursing, University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
No plan to share data. This was an instrument development study.

REFERENCES:
- [Result] Olson K, Rogers WT, Cui Y, Cree M, Baracos V, Rust T, Mellott I, Johnson L, Macmillan K, Bonville N. Development and psychometric testing of the Adaptive Capacity Index, an instrument to measure adaptive capacity in individuals with advanced cancer. Int J Nurs Stud. 2011 Aug;48(8):986-94. doi: 10.1016/j.ijnurstu.2011.01.013. Epub 2011 Feb 18. PMID 21333991